CLINICAL TRIAL: NCT04036240
Title: Finger Feeding as a Method of Human Milk Supplementation in Low Birth Weight Infants After Discharge: a Randomized Controlled Trial
Brief Title: Finger Feeding as a Method of HMF Supplementation After Discharge
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, YogaD, Head of Nutrition and Metabolic Diseases Division Dept of Child Health, Fakultas Kedokteran Universitas Indonesia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-05-0711
Record Dates: First submitted 2019-07-22; First posted 2019-07-29 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Low-Birth-Weight Infant; Breast Feeding
Keywords: low birth weight infant; breast milk supplementation; finger feeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Finger feeder (Experimental): HMF supplementation will be given by finger feeder
  Interventions: Other: Finger feeding
- Control (No Intervention): HMF supplementation will be given by mother preference such as cup, bottle.

INTERVENTIONS:
Other: Finger feeding — After discharge, subjects will be given HMF supplementation by finger feeding method using finger feeder
  Arms: Finger feeder

SUMMARY:
Human Milk Fortifier (HMF) is designed to supply additional calories, protein, vitamins and minerals to infants less than 37 weeks gestation or those less than 1500 g at birth. Liquid and powder types of HMF are available in the commercial market. Usually, one packet of powdered HMF is mixed to 25-50 cc expressed breast milk. Fortification of human milk is technically difficult in fully breastfed infants and artificial teats such as bottle feedings are common used. A study reported lower breastfeeding rate in intervention group who used HMF in comparison with control. Finger feeding method is associated with a better breastfeeding rate in hospital use. A feasibility study in Vienna reports finger feeding method as a way to provide fortification at home was acceptable.We hypothesize that finger feeding is an easy way for HMF supplementation after discharge to increase successful breastfeeding and improve growth in preterm and or low birth weight infants.

DETAILED DESCRIPTION:
For infants with very low birth weight (<1500 g) convincing evidence indicates that providing multi-nutrients fortification including protein, long-chain polyunsaturated fatty acid, and micro-nutrients improves infant growth during hospitalization and health outcomes. A study of predominantly breastfed preterm infants with fortification after discharge shows better growth than unsupplemented counterparts at 3 months corrected age. Another study showed that post discharged growth of < 1800 g infants with human milk fortifier (HMF) supplementation until 48 weeks gestational age improved. But without the intensive lactation counselling the breast milk in HMF group were lower than control group if artificial teats were used. 4. Finger feeding is an alternative method to feed infants to increase successful breastfeeding, but unpopular in Indonesia. Study on finger feeding are still limited and most study of them are not randomized trial. We evaluate the method of supplementation on breastfeeding rate, growth and safety. We also do in depth interview with those who have high or low compliance.

ELIGIBILITY:
Inclusion Criteria:

* birth weight < 2500 g
* need HMF supplementation after discharge
* predominantly breastfed
* live in Jakarta city and its surrounding
* parents agree to follow study procedure with signed informed consent

Exclusion Criteria:

* major congenital anomaly or other conditions interfere with normal growth and oral feeding

Min Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2019-07-22 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding rate | 28 days
  Formula used (ml/kg/day)

SECONDARY OUTCOMES:
Growth | 28 days
  mean difference in weight, length, head circumference; skin fol thickness (mm)
Compliance | 28 days
  Number of supplementation per day
Stool consistency | up to 1 month
  Diapered infant stool scale (1-5B)
Stool frequency | up to 1 month
  Number of stool per day
Vomiting | 4 weeks
  number per day
Choking | up to 1 month
  Number per day
Infections | up to 1 month
  Fever or other acute illness episode

OTHER OUTCOMES:
Mothers's opinion about finger feeder supplementation | up to 1 month
  In depth interview with guided questionnaire about using finger feeder at home (qualitative data)

CONTACTS AND LOCATIONS:
Overall Officials: Yoga Devaera, MD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (4):
- Indonesia (4):
  - Budi Kemuliaan Hospital, Jakarta Pusat, Jakarta Special Capital Region
  - RS Hermina Bekasi, Bekasi, West Java
  - RS Hermina Jatinegara, Jakarta
  - Koja District Hospital, Jakarta

IPD SHARING:
Plan to Share IPD: Yes
All IPD in results after publication
Supporting Information: Study Protocol
Time Frame: After publication
Access Criteria: systematic review proposal